CLINICAL TRIAL: NCT04441866
Title: Automated Analysis Algorithms in Second Trimester Obstetric Ultrasound
Acronym: Auto-2T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Federico Prefumo, Associate Professor, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NP3574
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Ultrasonography, Prenatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated algorithms (Active Comparator): Automated 3D techniques in measuring fetal biometry and reconstructing standard anatomical planes
  Interventions: Diagnostic Test: Automated algorithms
- Standard technique (Placebo Comparator): Standard 2D assessment
  Interventions: Diagnostic Test: Standard technique

INTERVENTIONS:
Diagnostic Test: Automated algorithms — Automated algorithms for measuring fetal biometry, and for the reconstruction of standard planes of fetal anatomy
  Arms: Automated algorithms
Diagnostic Test: Standard technique — Standard ultrasound examination without use of automated algorithms for measuring fetal biometry, and for the reconstruction of standard planes of fetal anatomy
  Arms: Standard technique

SUMMARY:
This study aims to evaluate the effect of the use of automated algorithms for the measurement of fetal biometry, and for the reconstruction of standard planes of fetal anatomy, compared with the standard ultrasound technique, during the second trimester ultrasound scan.

DETAILED DESCRIPTION:
In recent years in many ultrasound equipment were fitted with automated algorithms for measuring fetal biometry, and for the reconstruction of standard planes of fetal anatomy. Although there are studies that have assessed the application of these algorithms in terms of repeatability of the measurements made, or of possibility of acquiring diagnostic planes, there are no randomized controlled studies that evaluated their impact on the second trimester ultrasound scan.

The aim of the study is to evaluate the effect of the use of automated algorithms for the measurement of fetal biometry, and for the reconstruction of standard planes of fetal anatomy, compared with the standard ultrasound technique, in terms of:

* duration of the ultrasound scan
* quality of biometric measurements
* quality of the diagnostic planes
* operator satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy 19+0-21+6 weeks
* Live fetus
* No fetal abnormalities

Exclusion Criteria:

* Multiple pregnancy
* Intrauterine fetal death
* Fetal abnormalities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Duration of ultrasound examination | During ultrasound examination
  Duration of ultrasound examination in minutes

SECONDARY OUTCOMES:
Quality score of fetal biometry | During ultrasound examination
  Score described by Salomon et al. 2006: range from 0 (worst) to 16 (best)
Quality score of fetal diagnostic planes | During ultrasound examination
  Score described by Salomon et al. 2008: range from 0 (worst) to 32 (best)
Operator satisfaction | During ultrasound examination
  Visual analogue scale: from 0 (worst) to 32 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Spedali Ciivli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No